CLINICAL TRIAL: NCT07402148
Title: Research Proposal on the Effects of Different Altitude Conditions on Human Time Perception
Status: Not yet recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: KYLL-202503-033-2
Record Dates: First submitted 2025-11-27; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Heart Rate Monitoring
Keywords: different altitude conditions; vital signs; Time perception ability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: high-altitude environment — A high-altitude simulation chamber is used to simulate the environmental conditions at different altitudes

SUMMARY:
The aim of this observational study is to investigate human time perception ability for different time intervals (540 ms, 1080 ms, 1620 ms, 2160 ms, 5 s, 10 s, 20 s, 50 s) under conditions of varying altitudes (500 m, 1000 m, 1500 m, 2000 m, 2500 m, 3000 m). Specifically, a hypobaric chamber will be used to simulate the aforementioned altitudes, and temporal reproduction tasks with different standard durations will be conducted at each altitude. The time difference between the actual perceived duration and the target duration will be calculated to assess the level of time perception ability-with a smaller difference indicating stronger time perception ability.

At each altitude, participants' heart rate (HR) and oxygen saturation (SpO₂) will also be monitored to explore the correlation between physiological status and time perception ability under different altitude conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-50 years;
2. Not taking any medication during the monitoring period;
3. No history of anemia;
4. Have lived in plain area for a long time, and have no history of traveling in high altitude area in recent two months;
5. May want to live in plateau in the future
6. Voluntarily participate in the study and sign the informed consent.

Exclusion Criteria:

All subjects were excluded from claustrophobia, schizophrenia, affective disorder, mental retardation and other serious mental disorders as well as major physical and nervous system diseases, and had not taken psychotropic drugs

-

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study recruited healthy adult volunteers who met the inclusion and exclusion criteria in a university in Shandong Province
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2026-02-10 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Human time perception ability | six months
  The time difference between the actual duration used and the target duration when performing temporal reproduction of the target time interval.

SECONDARY OUTCOMES:
heart rate | six months
  The number of heartbeats per minute
oxygen saturation | six months
  The percentage of oxyhemoglobin (HbO₂) in the blood relative to the total concentration of all bindable hemoglobin (Hb + HbO₂)

CONTACTS AND LOCATIONS:
Overall Officials: Zhang min, Study Chair — Shandong University Qilu Hospital
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No